CLINICAL TRIAL: NCT07156643
Title: A Prospective, Single-arm, Multicenter Exploratory Clinical Study of Anlotinib Combined With Bempegaldesleukin and Conventional Chemoradiotherapy for the Treatment of Unresectable Locally Advanced or Metastatic Soft Tissue Sarcoma.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-485
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Soft Tissue Sarcoma
MeSH Terms: interventions — anlotinib; bempegaldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib in combination with bempegaldesleukin and conventional chemoradiotherapy (Experimental): Anlotinib in combination with bempegaldesleukin and conventional chemoradiotherapy
  Interventions: Drug: Anlotinib and bempegaldesleukin

INTERVENTIONS:
Drug: Anlotinib and bempegaldesleukin — Subjects will receive concurrent anlotinib, bempegaldesleukin, and radiotherapy, followed by maintenance therapy with anlotinib, bempegaldesleukin, and chemotherapy.
  Concurrent Radiotherapy Phase:
  Anlotinib: 10 mg orally once daily on days 1-14, every 3 weeks (q3w), for 2 cycles during radiotherapy.
  Bempegaldesleukin: 1200 mg IV on day 1, q3w, for 2 cycles during radiotherapy. Radiotherapy: Delivered once daily, with a total biological effective dose (BED) of 36-100 Gy. Techniques may include conventional fractionation or stereotactic body radiotherapy (SBRT), as determined by the investigator.
  Maintenance Phase:
  Chemotherapy: Doxorubicin 40 mg/m² IV day 1 + ifosfamide 1.2-2.4 g/m² IV days 1-5 per 21-day cycle for 4-6 cycles.
  Anlotinib: 10 mg orally once daily on days 1-14, q3w. Bempegaldesleukin: 1200 mg IV on day 1, q3w.

SUMMARY:
This study employs a multicenter, single-arm trial design. Participants will receive a treatment regimen consisting of "anlotinib plus bempegaldesleukin concurrent with radiotherapy," followed by a maintenance therapy phase of "anlotinib plus bempegaldesleukin concurrent with chemotherapy." The study aims to evaluate the clinical efficacy and safety of anlotinib in combination with bempegaldesleukin and conventional chemoradiotherapy for the treatment of unresectable locally advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
This multicenter, single-arm study is designed to enroll 46 patients with metastatic or unresectable locally advanced soft tissue sarcoma. Participants will receive a treatment regimen consisting of "anlotinib plus bempegaldesleukin concurrent with radiotherapy," followed by a maintenance phase of "anlotinib plus bempegaldesleukin concurrent with chemotherapy." The primary endpoint is objective response rate (ORR). Secondary endpoints include progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and safety. The study aims to evaluate the clinical efficacy and safety of anlotinib in combination with bempegaldesleukin and conventional chemoradiotherapy for the treatment of this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 80 years.
2. Diagnosis: Pathologically confirmed, investigator-assessed metastatic or unresectable locally advanced soft tissue sarcoma, classified as Stage IV according to the AJCC (8th Edition) staging system. Eligible histologic subtypes per the WHO (2013) classification include anthracycline-insensitive types, primarily: myxoid/round cell liposarcoma, Grade 1 dedifferentiated liposarcoma, clear cell sarcoma, endometrial stromal sarcoma, alveolar soft part sarcoma, extraskeletal myxoid chondrosarcoma, osteosarcoma, chondrosarcoma, Ewing sarcoma/primitive neuroectodermal tumor (PNET), embryonal rhabdomyosarcoma, alveolar rhabdomyosarcoma, gastrointestinal stromal tumor (GIST), etc. Eligibility of other rare soft tissue sarcoma subtypes will be determined by the investigator.
3. Measurable Disease: At least one measurable or evaluable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
4. Life Expectancy: ≥ 3 months.
5. Performance Status: Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
6. Adequate Organ Function: Must meet the following criteria within 7 days prior to treatment initiation:1）Hematological (without transfusion or use of growth factors within 14 days):Hemoglobin (Hb) ≥ 90 g/L,Absolute Neutrophil Count (ANC) ≥1.5 × 10⁹/L,Platelet count (PLT) ≥75×10⁹/L;Biochemical:Total Bilirubin (TBIL) ≤1.5 × Upper Limit of Normal (ULN),Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)≤ 2.5× ULN,Serum Creatinine (Cr)≤ 1.5 × ULN or Creatinine Clearance (CrCl) ≥ 60 mL/min,Urinalysis: Urine protein< 2+ and 24-hour urine protein quantification must show protein≤1 g;Coagulation: International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN;Cardiac Function: Left Ventricular Ejection Fraction (LVEF) ≥ 50% as assessed by Doppler ultrasound;Thyroid Function: Thyroid-Stimulating Hormone (TSH) ≤ 2.0 × ULN; if abnormal, T3 and T4 levels must be within normal limits for enrollment.
7. Contraception: Women of childbearing potential must have used reliable contraception, have a negative pregnancy test (serum or urine) within 7 days prior to enrollment, and be willing to use adequate contraception during the trial and for 8 weeks after the last dose of the study drug. Men must agree to use adequate contraception or be surgically sterile during the trial and for 8 weeks after the last dose.
8. Treatment Plan and Consent: The investigator plans to administer the combined chemoradiotherapy and targeted immunotherapy regimen, and the patient has provided written informed consent.

Exclusion Criteria:

1. Prior treatment with PD-1/PD-L1/CTLA-4 antibodies, radiotherapy, or any targeted therapy.
2. Tumor invasion of major blood vessels.
3. Active, known, or suspected autoimmune disease.
4. Known history of primary immunodeficiency.
5. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
6. Pregnant or lactating female patients.
7. Uncontrolled concurrent illnesses, including but not limited to:HIV infection (HIV antibody positive).Active or clinically poorly controlled severe infection.Active hepatitis.Evidence of severe or uncontrolled systemic diseases (e.g., severe psychiatric, neurological, epileptic, or dementia disorders; unstable or decompensated respiratory, cardiovascular, hepatic, or renal diseases; uncontrolled hypertension [defined as ≥ Grade 2 hypertension per CTCAE despite medical therapy]).Active bleeding or newly diagnosed thrombotic disease requiring therapeutic anticoagulation, or bleeding tendency; coagulation abnormalities (INR > 1.5 × ULN, APTT > 1.5 × ULN).
8. Current participation in another drug clinical trial.
9. Any other condition deemed by the investigator to make the patient unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Objective Response Rate (ORR) refers to the proportion of patients in whom tumor burden decreases by a predefined amount and remains reduced for a minimum time period. It encompasses both Complete Response (CR) and Partial Response (PR) cases. Tumor response is evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Progression-free Survival（PFS） | 2 years
  Progression-Free Survival (PFS) is defined as the time from the date of the first administration of the study drug to the date of disease progression or death from any cause, whichever occurs first.
Overall Survival（OS） | 2 years
  Overall Survival (OS) is defined as the time from the date of the first administration of the study drug to the date of death from any cause.
Disease control rate（DCR） | 2 years
  Disease Control Rate (DCR) refers to the proportion of patients in whom tumor burden decreases or remains stable according to predefined criteria, sustained for a minimum specified duration. It encompasses cases achieving Complete Response (CR), Partial Response (PR), and Stable Disease (SD). Tumor response is evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

OTHER OUTCOMES:
Number of Safety Events | 2 years
  Adverse Event and Adverse Drug Reaction and Serious Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No